CLINICAL TRIAL: NCT02351037
Title: A Multicenter Open-Label Phase 2a Study of Ibrutinib Monotherapy or in Combination With Either Cytarabine or Azacitidine in Subjects With Acute Myeloid Leukemia
Brief Title: Study of Ibrutinib in Subjects With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study data do not support development in AML.
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1131-CA
Record Dates: First submitted 2015-01-16; First posted 2015-01-30 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia; AML; Ibrutinib; Cytarabine; LD-AraC; Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ibrutinib; KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibrutinib Monotherapy Cohort (Experimental): Up to 33 response evaluable subjects will receive ibrutinib 560 mg once daily on a continuous basis.
  Interventions: Drug: Ibrutinib
- Ibrutinib + LD-AraC Combination Cohort (Experimental): Up to 25-28 additional response evaluable subjects (for a total of 34 subjects) will receive ibrutinib 560 mg once daily on a continuous basis starting 2 days prior to first cytarabine dose (20 mg BID sc) for 10 days of a 28-day cycle.
  Interventions: Drug: Ibrutinib + LD-AraC
- Ibrutinib+Azacitidine Combination Cohort (Experimental): Up to 34 response evaluable subjects will receive ibrutinib 560 mg once daily on a continuous basis starting 1 day prior to first azacitidine dose + azacitidine 75mg/m2 IV once daily Days 1-7 of a 28-day cycle (with an option to increase to 100mg/m2 after 2 cycles).
  Interventions: Drug: Ibrutinib+Azacitidine

INTERVENTIONS:
Drug: Ibrutinib — Subjects will receive ibrutinib 560 mg once daily on a continuing basis.
  Other Names: Cohort 1
  Arms: Ibrutinib Monotherapy Cohort
Drug: Ibrutinib + LD-AraC — Subjects will receive ibrutinib 560 mg once daily on a continuous basis starting 2 days prior to first cytarabine dose (20 mg BID sc) for 10 days of a 28-day cycle.
  Other Names: Cohort 2
  Arms: Ibrutinib + LD-AraC Combination Cohort
Drug: Ibrutinib+Azacitidine — Subjects will receive ibrutinib 560 mg once daily on a continuous basis starting 1 day prior to first azacitidine dose + azacitidine 75 mg/m2 IV once daily on Days 1-7 of a 28-day cycle (with an option to increase to 100 mg/m2 after 2 cycles).
  Other Names: Cohort 3
  Arms: Ibrutinib+Azacitidine Combination Cohort

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of ibrutinib alone or in combination with either cytarabine or azacitidine in the treatment of subjects with Acute Myeloid Leukemia (AML) who have failed standard treatment, or subjects without prior therapy who refuse standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subjects with pathologically documented AML that has failed standard treatment, or subjects without prior therapy who refuse standard treatment options
* Bone marrow aspirate/biopsy results showing >5% blasts
* WBC count <25,000 cells/mm3 (25 x 109/L)
* Platelet count >10,000 cells/mm3 (10 x 109/L)
* Adequate hepatic and renal function defined as:

  * For Cohorts 1 and 2: serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤3.0 x upper limit of normal (ULN); for Cohort 3: ALT ≤2.5 or AST ≤2.5 ULN.
  * Serum creatinine ≤2 mg/dL or Estimated Creatinine Clearance ≥30 mL/min (Cockcroft-Gault).
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
* PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN (When treated with warfarin or other vitamin K antagonists, then INR ≤3.0).
* Female subjects who are of non-reproductive potential (Female subjects of reproductive potential must have a negative serum pregnancy test upon study entry).
* Male and female subjects of reproductive potential agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) during the period of therapy and for 90 days after the last dose of study drug.

Exclusion Criteria:

* Acute promyelocytic leukemia (French-American-British Class M3 AML).
* Known active central nervous system (CNS) leukemia.
* Known active systemic infection (Grade ≥2).
* Active bleeding disorders or clinical signs of bleeding (Grade ≥2).
* Prior bone marrow transplant that requires immunosuppressant therapy or presents with graft vs host disease (GVHD).
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and with low risk of recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* Prior treatment with a BTK inhibitor.
* For Cohort 3 subjects, prior treatment with hypomethylating agents (eg, azacitidine, decitabine)
* Anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal or any investigational therapy within 14 days or 5 half-lives (whichever is shorter) prior to first dose of study drug.
* Subject has received a monoclonal antibody for anticancer intent within 8 weeks prior to the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring intravenous (IV) systemic treatment that was completed ≤14 days before the first dose of study drug.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), Grade 0 or 1, unless otherwise defined in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Major surgery within 4 weeks of first dose of study drug.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Concomitant use of warfarin or other Vitamin K antagonists.
* Requires treatment or prophylaxis with a strong cytochrome P450 (CYP) 3A inhibitor
* Currently active, clinically significant hepatic impairment (≥ moderate hepatic impairment according to the Child Pugh classification).
* Lactating or pregnant.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - UC Davis Medical Center, Sacramento, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Einstein Center for Cancer Research, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilken R, Li CS, Sharon VR, Kim K, Patel FB, Patel F, Maverakis E. Topical clobetasol for the treatment of toxic epidermal necrolysis: study protocol for a randomized controlled trial. Trials. 2015 Aug 22;16:374. doi: 10.1186/s13063-015-0879-7. PMID 26297574

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibrutinib Monotherapy Cohort | Ibrutinib + LD-AraC Combination Cohort | Ibrutinib+Azacitidine Combination Cohort
Started | 7 | 21 | 8
Completed | 7 | 21 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib Monotherapy Cohort | Ibrutinib + LD-AraC Combination Cohort | Ibrutinib+Azacitidine Combination Cohort | Total
Number analyzed (Participants) | 7 | 21 | 8 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 6 | 15
  >=65 years | 3 | 16 | 2 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11.7) | 70 (9.1) | 58 (12.4) | 67 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 6 | 16
  Male | 4 | 14 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 6 | 19 | 6 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 6 | 19 | 8 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 21 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Ibrutinib Monotherapy or in Combination With Either LD-AraC or Azacitidine Using the Overall Remission Rate (Defined as Proportion of Subjects Achieving a CR or CRi) According to the LeukemiaNet Guidelines
Description: Dohner's 2000 Criteria for AML: Complete Response (CR), Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100 000/µL); independence of red cell transfusions; CR with Incomplete Recovery (CRi), All CR criteria except for residual neutropenia (< 1.0 x 109/L [1000/µL]) or thrombocytopenia (<100 x 109/L [100 000/µL]) ; Morphologic leukemia-free state, Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required; Partial Remission (PR), All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%; Relapse, Bone marrow blasts > 5%; or reappearance of blasts in the blood; or development of extramedullary disease.
Time Frame: When the last subject enrolled completes approximately 12 months of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib Monotherapy Cohort | Ibrutinib + LD-AraC Combination Cohort | Ibrutinib+Azacitidine Combination Cohort
Number analyzed (Participants) | 7 | 21 | 8
Participants | 0 | 1 | 0

2. Primary Outcome: Safety and Tolerability of Ibrutinib Monotherapy or in Combination With Either LD-AraC or Azacitidine
Description: Number of Participants with Adverse Events and number of patients with lab abnormalities.The safety profile of ibrutinib was evaluated based on the incidence of adverse events (AEs) as well as clinically significant laboratory abnormalities and vital signs, and other malignancies. The safety evaluations performed in this study were standard and/or were required based on the safety data available from other clinical and preclinical settings.
Time Frame: Up to 30 days following the last dose of study drug.
Reporting Status: Not Posted

3. Secondary Outcome: Relapse-free Survival (RFS), Event-free Survival (EFS) and Overall Survival (OS)
Description: To evaluate clinical efficacy by assessing relapse-free survival (RFS), event-free survival (EFS) and overall survival (OS).
Time Frame: When the last subject enrolled completes approximately 12 months of treatment
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Benefit Rate - as Defined as the Proportion of Subjects Who Achieve CR, CRi, Morphologic Leukemia-free State, or Partial Remission (PR)
Description: To evaluate clinical benefit defined as CR, CRi, morphologic leukemia-free state, and partial remission (PR).
Time Frame: When the last subject enrolled completes approximately 12 months of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Arm/Group | Ibrutinib Monotherapy Cohort | Ibrutinib + LD-AraC Combination Cohort | Ibrutinib+Azacitidine Combination Cohort
All-Cause Mortality (participants affected / at risk) | 7/7 | 21/21 | 8/8
Serious Adverse Events (participants affected / at risk) | 4/7 | 21/21 | 8/8
Other Adverse Events (participants affected / at risk) | 7/7 | 21/21 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib Monotherapy Cohort (N=7) | Ibrutinib + LD-AraC Combination Cohort (N=21) | Ibrutinib+Azacitidine Combination Cohort (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 8 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Septic embolus (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 9 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib Monotherapy Cohort (N=7) | Ibrutinib + LD-AraC Combination Cohort (N=21) | Ibrutinib+Azacitidine Combination Cohort (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 5
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 2
Vision blurred (Eye disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 10 | 3
Nausea (Gastrointestinal disorders) | 3 | 8 | 3
Constipation (Gastrointestinal disorders) | 0 | 6 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 12 | 2
Oedema peripheral (General disorders) | 3 | 10 | 3
Pyrexia (General disorders) | 1 | 6 | 2
Asthenia (General disorders) | 0 | 7 | 0
Chills (General disorders) | 0 | 5 | 3
Malaise (General disorders) | 0 | 2 | 2
Injection site bruising (General disorders) | 1 | 2 | 0
Pain (General disorders) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 5 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 11 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 7 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 2
Headache (Nervous system disorders) | 2 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 5 | 1
Agitation (Psychiatric disorders) | 0 | 4 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 6 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Catheter site erythema (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Mass (General disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Granulicatella infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory fungal infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral sepsis (Infections and infestations) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access site occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema multiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until after the completion of the study or until 12 months after results are received

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT02351037/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02351037/SAP_001.pdf